CLINICAL TRIAL: NCT00517127
Title: A Comparison of Crystalloids vs. Colloids for Intraoperative Goal-directed Fluid Management
Brief Title: Crystalloids Versus Colloids During Surgery
Acronym: CC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Fresenius Kabi (Industry)
Responsible Party: Principal Investigator, Barbara Kabon, MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 431/2005
Record Dates: First submitted 2007-08-15; First posted 2007-08-16 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Fluid Overload; Postoperative Complications
Keywords: Intraoperative care; Ringer's lactate; Voluven; Cardiovascular diagnostic technique; Doppler effect
MeSH Terms: conditions — Edema; Postoperative Complications | interventions — Ringer's Lactate; Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Arm Nr 1: If corrected flow time (fTc), measured by esophageal doppler, falls below 350 msec, 250 ml of Lactated Ringer's Solution will be administered.
  Interventions: Drug: Lactated Ringer's Solution
- 2 (Active Comparator): Arm Nr 2: If corrected flow time (fTc), measured by esophageal doppler, falls below 350 msec, 250 ml of Hydroxyethylstarch 6% 130/0.4 will be administered.
  Interventions: Drug: Hydroxyethylstarch 6% 130/0.4

INTERVENTIONS:
Drug: Lactated Ringer's Solution — Arm Nr 1: If corrected flow time (fTc), measured by esophageal doppler, falls below 350 msec, 250 ml of Lactated Ringer's Solution will be administered.
  Arms: 1
Drug: Hydroxyethylstarch 6% 130/0.4 — Arm Nr 2: If corrected flow time (fTc), measured by esophageal doppler, falls below 350 msec, 250 ml of Hydroxyethylstarch 6% 130/0.4 will be administered.
  Arms: 2

SUMMARY:
The purpose of the study is to test whether colloid-based goal-directed intraoperative fluid management leads to less perioperative morbidity compared to crystalloid-based goal-directed intraoperative fluid management. Goal-directed therapy is based on measurements by an Esophageal Doppler Device.

DETAILED DESCRIPTION:
For a long time there is a raging debate whether crystalloid solutions or colloid solutions are better suited for fluid therapy. Early proponents both for crystalloids [Shires 1961] and colloids [Shoemaker 1979] deserve credit for elucidating important facts about volume replacement therapy - without answering the primary question. Elaborate reviews comparing crystalloid and colloid therapy for critically ill patients have been performed in the late nineties and updated recently [Roberts 2004]. However, it has been suggested that both questions and answers of reviews leave us none but wiser [Webb 1999]. Although a plethora of studies comparing crystalloid vs. colloid therapy in the last decades have been published, volume replacement therapy is still considered to be based on dogma and personal beliefs [Boldt 2003].

Goal-directed intraoperative fluid therapy monitored by Esophageal Doppler identifies volume-responders, thereby decreasing length of stay in hospital in orthopedic [Sinclair 1997], cardiac [Mythen 1995], and abdominal surgery patients [Gan 2002, Wakeling 2005, Noblett 2006]. However, all these studies have been performed with a colloid to be the substance applied. Thus, it has been questioned whether monitoring with the Esophageal Doppler monitor, or the application of additional colloid improved outcome [Horowitz, Kumar 2003].

Consequently, the researchers will use Esophageal Doppler Monitoring for intraoperative goal-directed fluid therapy to compare the effects of crystalloid vs. colloid therapy on various organ systems, assessing combined perioperative morbidity [Bennett-Guerrero 1999] .

ELIGIBILITY:
Inclusion Criteria:

* After written informed consent patients undergoing elective open colon surgery, or open hysterectomy or myomectomy, or spine surgery or hip replacement will be included in the study.

Exclusion Criteria:

* Patients having severe cardiac or renal insufficiency
* Patients with severe coronary artery disease
* Patients with insulin-dependent diabetes mellitus
* Patients with severe COPD
* Patients with symptoms of infections or sepsis
* Patients with allergy to hydroxyethylstarch.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1109 (Actual)
Dates: Start 2006-09; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
combined perioperative morbidity | 30 days after surgery

SECONDARY OUTCOMES:
Tissue oxygenation, Wound Infection, Incidence of postoperative nausea and vomiting (PONV) and pain, pulmonary function, | 30 days after surgery

OTHER OUTCOMES:
Coagulation (ROTEM) | intraop, postop day1
  in a subgroup of 50 patients undergoing hepatic resection ROTEM measurements will be performed intraoperatively, postoperatively and on the first postoperative morning and compared between the groups.
Inflammatory response attenuation by HES 130/0.4 | 4 postoperative days
  In a subgroups of 120 patients the postoperative immune function will be evaluated and compared between crystalloids and colloids.
  The immunological parameters include:
  IL6, IL-8, IL-10, Procalcitonin, lipopolysaccharide-binding protein, HLA-DR Expression, CRP C-reactive protein, leucocytes, TNF alpha Blood samples will be collected immediately before surgery (T0) for baseline measurement, immediately after surgery finish (T1), and on postoperative day one, two and four (T2, T3 and T4).
Body Composition Monitor Measurement (BCM) | pre and postoperatively
  In a subgroup of 100 patients overhydration will be evaluated pre- and immediately postoperatively with a body composition monitor (BCM), a whole-body bioimpedance spectroscopy device manufactured and distributed by Fresenius Medical Care, Germany.
  Measurements will be compared betwwen the groups

CONTACTS AND LOCATIONS:
Overall Officials: Edith Fleischmann, M.D., Ph.D., Principal Investigator — Department of Anesthesiology, University of Vienna Medical School, Vienna, Austria
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Background] SHIRES T, WILLIAMS J, BROWN F. Acute change in extracellular fluids associated with major surgical procedures. Ann Surg. 1961 Nov;154(5):803-10. doi: 10.1097/00000658-196111000-00005. No abstract available. PMID 13912109
- [Background] Shoemaker WC, Hauser CJ. Critique of crystalloid versus colloid therapy in shock and shock lung. Crit Care Med. 1979 Mar;7(3):117-24. doi: 10.1097/00003246-197903000-00007. No abstract available. PMID 436427
- [Background] Roberts I, Alderson P, Bunn F, Chinnock P, Ker K, Schierhout G. Colloids versus crystalloids for fluid resuscitation in critically ill patients. Cochrane Database Syst Rev. 2004 Oct 18;(4):CD000567. doi: 10.1002/14651858.CD000567.pub2. PMID 15495001
- [Background] Webb AR. Crystalloid or colloid for resuscitation. Are we any the wiser? Crit Care. 1999;3(3):R25-R28. doi: 10.1186/cc346. No abstract available. PMID 11094479
- [Background] Boldt J. New light on intravascular volume replacement regimens: what did we learn from the past three years? Anesth Analg. 2003 Dec;97(6):1595-1604. doi: 10.1213/01.ANE.0000089961.15975.78. PMID 14633526 (Retraction: PMID 33031689 Anesth Analg. 2020 Aug;131(2):e137)
- [Background] Sinclair S, James S, Singer M. Intraoperative intravascular volume optimisation and length of hospital stay after repair of proximal femoral fracture: randomised controlled trial. BMJ. 1997 Oct 11;315(7113):909-12. doi: 10.1136/bmj.315.7113.909. PMID 9361539
- [Background] Mythen MG, Webb AR. Perioperative plasma volume expansion reduces the incidence of gut mucosal hypoperfusion during cardiac surgery. Arch Surg. 1995 Apr;130(4):423-9. doi: 10.1001/archsurg.1995.01430040085019. PMID 7535996
- [Background] Gan TJ, Soppitt A, Maroof M, el-Moalem H, Robertson KM, Moretti E, Dwane P, Glass PS. Goal-directed intraoperative fluid administration reduces length of hospital stay after major surgery. Anesthesiology. 2002 Oct;97(4):820-6. doi: 10.1097/00000542-200210000-00012. PMID 12357146
- [Background] Wakeling HG, McFall MR, Jenkins CS, Woods WG, Miles WF, Barclay GR, Fleming SC. Intraoperative oesophageal Doppler guided fluid management shortens postoperative hospital stay after major bowel surgery. Br J Anaesth. 2005 Nov;95(5):634-42. doi: 10.1093/bja/aei223. Epub 2005 Sep 9. PMID 16155038
- [Background] Noblett SE, Snowden CP, Shenton BK, Horgan AF. Randomized clinical trial assessing the effect of Doppler-optimized fluid management on outcome after elective colorectal resection. Br J Surg. 2006 Sep;93(9):1069-76. doi: 10.1002/bjs.5454. PMID 16888706
- [Background] Horowitz PE, Kumar A. It's the colloid, not the esophageal Doppler monitor. Anesthesiology. 2003 Jul;99(1):238-9; author reply 239. doi: 10.1097/00000542-200307000-00045. No abstract available. PMID 12826872
- [Background] Bennett-Guerrero E, Welsby I, Dunn TJ, Young LR, Wahl TA, Diers TL, Phillips-Bute BG, Newman MF, Mythen MG. The use of a postoperative morbidity survey to evaluate patients with prolonged hospitalization after routine, moderate-risk, elective surgery. Anesth Analg. 1999 Aug;89(2):514-9. doi: 10.1097/00000539-199908000-00050. PMID 10439777
- [Derived] Obradovic M, Luf F, Reiterer C, Schoppmann S, Kurz A, Fleischmann E, Kabon B. The effect of goal-directed crystalloid versus colloid administration on postoperative spirometry parameters: a substudy of a randomized controlled clinical trial. Perioper Med (Lond). 2024 Apr 15;13(1):28. doi: 10.1186/s13741-024-00381-z. PMID 38622671
- [Derived] Obradovic M, Kurz A, Kabon B, Roth G, Kimberger O, Zotti O, Bayoumi A, Reiterer C, Stift A, Fleischmann E. The effect of intraoperative goal-directed crystalloid versus colloid administration on perioperative inflammatory markers - a substudy of a randomized controlled trial. BMC Anesthesiol. 2020 Aug 21;20(1):210. doi: 10.1186/s12871-020-01126-3. PMID 32825817
- [Derived] Reiterer C, Kabon B, Zotti O, Obradovic M, Kurz A, Fleischmann E. Effect of goal-directed crystalloid- versus colloid-based fluid strategy on tissue oxygen tension: a randomised controlled trial. Br J Anaesth. 2019 Dec;123(6):768-776. doi: 10.1016/j.bja.2019.08.027. Epub 2019 Oct 15. PMID 31627889